CLINICAL TRIAL: NCT07367204
Title: A Prospective, Multicenter, Randomized, Parallel-Controlled, Subject- and Investigator-Masked, Non-Inferiority Clinical Trial to Evaluate the Efficacy and Safety of Cross-Linked Hyaluronic Acid Gel for Injection in Correcting Moderate to Severe Nasolabial Folds
Brief Title: Randomized Masked Trial of Injectable Cross-Linked Hyaluronic Acid for Moderate-to-Severe Nasolabial Folds
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing Jinsaixing Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-OM003-PCT01
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Nasolabial Fold Wrinkles
MeSH Terms: interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subject-Blinded, Evaluator-Blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intense (Experimental)
  Interventions: Device: Intense
- Restylane (Active Comparator)
  Interventions: Device: Restylane

INTERVENTIONS:
Device: Intense — Correction of moderate to severe nasolabial fold wrinkles
  Arms: Intense
Device: Restylane — the Correction of Midface Volume Deficiency and/or Midface Contour Deficiency
  Arms: Restylane

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of injectable cross - linked hyaluronic acid gel for correcting moderate to severe nasolabial fold wrinkles, on the premise of ensuring the safety of subjects and the scientific rigor of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 26 years (inclusive), regardless of gender;
2. Subjects willing to correct nasolabial fold wrinkles;
3. Subjects with bilateral nasolabial folds having the same WSRS grade (both Grade 3 or both Grade 4) as assessed by masked evaluators;
4. Subjects who can understand the purpose of the study, voluntarily participate, and are willing to sign a written informed consent form.

Exclusion Criteria:

1. Subjects with known allergies to hyaluronic acid products or any components of the investigational medical device/control medical device; or subjects with a known history of severe allergies or anaphylactic shock;
2. Subjects with abnormal coagulation function at screening (Activated Partial Thromboplastin Time [APTT] > 1.5 × upper limit of normal [ULN]), or those who have used any thrombolytics, anticoagulants, or antiplatelet drugs (e.g., warfarin, aspirin, etc.) within 2 weeks prior to screening;
3. Presence of tattoos, piercings, significant facial hair, scars, deformities, unhealed wounds, abscesses, granulomas, active or persistent perinasal infections, malignancies or precancerous lesions, malignant tumors, or skin masses of unknown nature in the injection area and adjacent sites that may affect efficacy assessment or increase treatment risks;
4. Presence of active skin diseases, inflammation, or infections (e.g., herpes, acne, eczema, dermatitis, psoriasis, shingles, mycosis, papilloma, etc.) that, in the investigator's judgment, may affect efficacy assessment or increase treatment risks;
5. Subjects who have received or plan to receive surgical treatments for facial wrinkle improvement (e.g., autologous fat transplantation, absorbable suture embedding therapy, or facelift surgery) in the injection area and adjacent sites within 12 months prior to screening or during the study, which, in the investigator's judgment, may affect efficacy assessment or increase treatment risks;
6. Subjects who have received or plan to receive injections of any permanent fillers (e.g., polymethylmethacrylate [PMMA], silicone, expanded polytetrafluoroethylene [ePTFE], etc.) or other unknown materials in the injection area and adjacent sites;
7. Subjects who have received or plan to receive treatments with calcium hydroxylapatite, poly-L-lactic acid [PLLA], polylactic acid, poly-DL-lactic acid [PDLLA], polycaprolactone [PCL], etc., in the injection area and adjacent sites within 24 months prior to screening or during the study;
8. Subjects who have received or plan to receive cross-linked sodium hyaluronate injection therapy in the injection area and adjacent sites within 12 months prior to screening or during the study;
9. Subjects who have received or plan to receive any cosmetic treatments or facial surgeries (e.g., botulinum toxin therapy, non-cross-linked sodium hyaluronate filling, collagen filling, radiofrequency therapy, focused ultrasound therapy, intense pulsed light [IPL], laser therapy, medium or deeper chemical peels, dermabrasion, liposuction, fat dissolution, photodynamic therapy, or other ablative surgeries, etc. [excluding mesotherapy]) in the injection area and adjacent sites within 6 months prior to screening or during the study;
10. Subjects who have received or plan to receive mesotherapy, photobiomodulation (e.g., red and blue light, excluding laser therapy), intense pulsed light, microneedling (excluding radiofrequency microneedling), or very superficial or superficial chemical peels (e.g., retinol, alpha-hydroxy acids [AHAs], salicylic acid, etc.) in the injection area and adjacent sites within 3 months prior to screening or during the study;
11. Subjects with active autoimmune diseases (e.g., inflammatory bowel disease) or a history thereof, or active connective tissue diseases (e.g., rheumatoid arthritis, scleroderma, and systemic lupus erythematosus) or a history thereof;
12. Subjects who have received chemotherapy, immunosuppressant therapy, immunomodulator therapy (e.g., monoclonal antibodies, etc.), or systemic corticosteroid therapy (excluding inhaled corticosteroids) within 3 months prior to screening; or those who have taken retinoids within 6 months prior to screening; or those who have received any drug therapy within 1 month prior to screening or within 5 drug half-lives (whichever is longer), which, in the investigator's judgment, may affect efficacy assessment or increase treatment risks;
13. Subjects with a history of keloid formation, tendency to develop hypertrophic scars, or any other healing disorders;
14. Subjects with significant facial edema or diseases expected to cause facial edema during the study, which, in the investigator's judgment, may affect injection safety or efficacy assessment;
15. Subjects with severe impairment of major organ function (brain, heart, lungs, liver, kidneys, etc.) as judged by the investigator, such as severe cardiovascular and cerebrovascular diseases (hospitalization for myocardial infarction or cardiac surgery within 3 months, history of congestive heart failure or myocardial infarction, severe unstable arrhythmia, hypertrophic cardiomyopathy, severe aortic stenosis, aneurysm, stroke, etc.), severe pulmonary diseases (moderate to severe pneumonia, respiratory failure, etc.), uncontrolled diabetes mellitus, epilepsy, or history of severe mental illness, psychological disorders, visual impairment, etc.;
16. Subjects with full dentures or any devices covering all or part of the palate, severe malocclusion, dental or maxillofacial deformities, or significant perioral asymmetry, which, in the investigator's judgment, may affect efficacy assessment or increase treatment risks;
17. Subjects who have received or plan to receive dental treatments that may affect efficacy assessment (e.g., tooth extraction, orthodontic treatment, dental implants, etc.) within 3 months prior to screening or during the study;
18. Subjects planning to have a significant weight change (>10% body weight change) during the clinical trial;
19. Female subjects who are pregnant, lactating, or planning to conceive during the clinical trial;
20. Subjects currently participating in other clinical trials, or those who participated in a drug clinical trial within 3 months, or a medical device clinical trial within 1 month (excluding cases where only informed consent was signed without receiving any intervention);
21. Other conditions deemed inappropriate for participation in the study by the investigator.

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2027-03-06 (Estimated)

PRIMARY OUTCOMES:
Effective rate of nasolabial fold wrinkle improvement at 180 ± 14 days after the last injection (assessed by masked evaluators). | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China